CLINICAL TRIAL: NCT07069673
Title: Abbott Cephea Mitral Valve Disease Registry
Status: Recruiting | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: ABT-CIP-10593
Record Dates: First submitted 2025-06-23; First posted 2025-07-17 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-10

CONDITIONS: Mitral Regurgitation; Mitral Stenosis; Mitral Valve Disease; Mitral Valve (MV) Regurgitation; Mitral Annulus Calcification; Mitral Valve Replacement; Transcatheter Valve Replacement
Keywords: Mitral Valve Disease; registry; Cephea Mitral Valve System
MeSH Terms: conditions — Mitral Valve Insufficiency; Mitral Valve Stenosis; Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Potential transcatheter mitral valve replacement (TMVR) candidates: Patients with symptomatic mitral valve disease who may be candidates for transcatheter mitral valve replacement.

SUMMARY:
The objective of this registry is to gather clinical data on symptomatic patients with mitral valve disease, including patients with mitral regurgitation, mitral stenosis, and mixed mitral valve disease. Data collected from this registry are expected to improve our understanding of the impact of correcting symptomatic mitral valve disease on clinical outcomes in patients that could be candidates for Transcatheter Mitral Valve Replacement and may also inform future regulatory or reimbursement submission strategies for the Cephea Mitral Valve System.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic mitral valve disease resulting in mitral regurgitation and/or severe mitral valve stenosis.
2. New York Heart Association (NYHA) Functional Class II, III, or ambulatory IV.
3. In the judgement of the Site Heart Team, transcatheter therapy is deemed to be more appropriate than conventional mitral valve surgery, TMVR is more likely to provide an optimal result than TEER, and the subject has been adequately treated per applicable standards, including for coronary artery disease, left ventricular dysfunction, and heart failure.
4. Age 18 years or older at time of consent.
5. The subject agrees to the study requirements, permits all follow-up data entry, and has provided written informed consent.

Exclusion Criteria:

1. Prior surgical or interventional treatment that interferes with the Cephea valve delivery or function.
2. Subject is undergoing dialysis or experiencing chronic renal failure
3. Subject has chronic lung disease requiring continuous home oxygen therapy or chronic outpatient oral steroid use
4. Subjects with comorbidities that are likely to result in a life expectancy of less than 12 months.
5. Pregnant or nursing subjects and those who plan pregnancy during the follow-up period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This registry will enroll subjects over 18 years of age of all genders with symptomatic mitral valve disease including those with mitral regurgitation, mitral stenosis, and mixed mitral valve disease, who are candidates for transcatheter mitral valve replacement.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-08-13 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Primary Objective | From enrollment to 2 years of follow-up
  The objective of the MVD Registry is to collect data on the progression of MVD patients considered for TMVR therapy to guide product development, regulatory submissions, and reimbursement planning

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Phoenix Cardiovascular Research Group, Phoenix, Arizona
  - Los Robles Regional Medical Center, Thousand Oaks, California
  - Piedmont Heart Institute, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Ascension St. Vincent, Indianapolis, Indiana
  - Via Christi Regional Medical Center - St. Francis Campus, Wichita, Kansas
  - Providence St. Patrick Hospital, Missoula, Montana
  - Allegheny General Hospital - ASRI, Pittsburgh, Pennsylvania
  - TriStar Centennial Medical Center, Nashville, Tennessee
  - Ascension Saint Thomas, Nashville, Tennessee
  - Vanderbilt Heart & Vascular Institute, Nashville, Tennessee
  - Houston Methodist, Houston, Texas
  - UTHealth Memorial Hermann, Houston, Texas
  - Sentara Norfolk General Hospital, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No